CLINICAL TRIAL: NCT03661528
Title: A Randomized Clinical Trial of Andexanet Alfa in Acute Intracranial Hemorrhage in Patients Receiving an Oral Factor Xa Inhibitor
Brief Title: Trial of Andexanet Alfa in ICrH Patients Receiving an Oral FXa Inhibitor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-513; 2018-002620-17 (EudraCT Number)
Record Dates: First submitted 2018-08-30; First posted 2018-09-07 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Acute Intracranial Hemorrhage
Keywords: thrombosis; anticoagulant; acute intracranial hemorrhage; andexanet alfa
MeSH Terms: conditions — Thrombosis | interventions — PRT064445

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: ANNEXA-I is a randomized, open-label study with blinded adjudication on primary efficacy and safety outcomes, including death and thrombotic events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- andexanet alfa (Experimental): Patients will receive one of two dosing regimens of andexanet alfa based on which FXa inhibitor they received and the amount and timing of the most recent dose.
  Interventions: Drug: andexanet alfa
- Usual Care (Other): Usual care will consist of any treatment(s) (including no treatment) other than andexanet alfa administered within 3 hours post-randomization that the Investigator and/or other treating physicians consider to be appropriate.
  Interventions: Drug: Usual Care

INTERVENTIONS:
Drug: andexanet alfa — Andexanet alfa is a recombinant version of human FXa
  Arms: andexanet alfa
Drug: Usual Care — Usual care will consist of any treatment(s) (including no treatment) other than andexanet alfa administered within 3 hours post-randomization that the Investigator and/or other treating physicians consider to be appropriate.
  Arms: Usual Care

SUMMARY:
Randomized, controlled clinical trial evaluating the efficacy and safety of andexanet alfa versus usual care in patients with intracranial hemorrhage anticoagulated with a direct oral FXa anticoagulant

DETAILED DESCRIPTION:
This is a randomized, multicenter clinical trial designed to determine the efficacy and safety of andexanet alfa compared to usual care in patients presenting with acute intracranial hemorrhage within 6 hours of symptom onset to baseline scan and within 15 hours of taking an oral factor Xa inhibitor. The study will use a prospective, randomized, open label (PROBE) design. The primary efficacy outcome will be adjudicated by a blinded Endpoint Adjudication Committee. To support the adjudication of hemostatic efficacy, a blinded Imaging Core Laboratory will review all available scans. Between 900 and 1200 patients are planned to be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent. Either the patient or his or her medical proxy (or legally authorized representative if permissible by local or regional laws and regulations) has been adequately informed of the nature and risks of the study and has given written informed consent prior to Screening.

   * Deferred consent procedure is allowed where approved by local ethics committees. In cases of deferred consent, the time of the study physician's documented decision to include the patient into the study will serve as "time of consent" with respect to protocol-specific procedures.
   * In all cases where the patient does not sign informed consent prior to study entry, informed consent from the patient will be obtained as soon as realistically possible after inclusion in the trial and in accordance with the Declaration of Helsinki, International Conference on Harmonization-Good Clinical Practice (GCP), the EU General Data Protection Regulation (GDPR) and national and local regulations.
2. Age ≥ 18 years old at the time of consent.
3. An acute intracerebral bleeding episode, defined as an estimated blood volume ≥ 0.5 to ≤ 60 mL acutely observed radiographically within the cerebrum. Patients may have extracerebral (e.g., subdural, subarachnoid, epidural) or extracranial (e.g., gastrointestinal, intraspinal) bleeding additionally, but the intracerebral hemorrhage must be considered the most clinically significant bleed at the time of enrollment.
4. Performance of a head CT or MRI scan demonstrating the intracerebral bleeding within 2 hours prior to randomization (the baseline scan may be repeated only once to meet this criterion).
5. Treatment with an oral FXa inhibitor (apixaban [last dose 2.5 mg or greater], rivaroxaban [last dose 10 mg or greater], or edoxaban [last dose 30 mg or greater]):

   * ≤ 15 hours prior to randomization.
   * > 15 hours prior to randomization or unknown time of last dose, if documented anti fXa activity is > 100 ng/mL for direct fXa inhibitors (apixaban, rivaroxaban or edoxaban) may be enrolled, irrespective of the time of the last dose, and the local anti-fXa activity level is obtained within 2 hours prior to consent, performed as per standard of care. Note: Patients enrolled in this manner should receive a high andexanet dosing regimen.
6. Time from bleeding symptom onset < 6 hours prior to the baseline imaging scan. Time of trauma (if applicable) or time last seen normal may be used as surrogates for time of symptom onset. (If the baseline scan is repeated to meet Inclusion Criterion #4, the time from bleeding symptom onset must be < 6 hours prior to the repeat baseline imaging scan.)
7. Female patients of childbearing potential and male patients with female partners of childbearing potential must follow protocol-specified guidance for avoiding pregnancy for 30 days after the last dose of study drug.
8. Have a negative pregnancy test documented prior to enrollment (for females of childbearing potential).
9. NIHSS score ≤ 35 at the time of consent.

Exclusion Criteria

If a patient meets any of the following criteria, he or she is not eligible to participate in this trial:

1. Planned surgery, including Burr holes for hematoma drainage, within 12 hours after randomization. Minimally invasive surgery/procedures not directly related to the treatment of intracranial bleeding and that are not expected to significantly affect hematoma volume are allowed (e.g., Burr holes for intracranial pressure monitoring, endoscopy, bronchoscopy, central lines.
2. GCS score < 7 at the time of consent. If a patient is intubated and/or sedated at the time of consent, they may be enrolled if it can be documented that they were intubated/sedated for non-neurologic reasons within 2 hours prior to consent.
3. Purposefully left blank.
4. Anticipation that the baseline and follow up brain scans will not be able to use the same imaging modalities (i.e., patients with a baseline CT scan should have a CT scan in follow up; similarly, for MRI).
5. Expected survival of less than 1 month (not related to the intracranial bleed).
6. Recent history (within 2 weeks) of a diagnosed TE or clinically relevant symptoms of the following:

   ○ Venous Thromboembolism (VTE: e.g., deep venous thrombosis, PE, cerebral venous thrombosis), myocardial infarction (MI), Disseminated Intravascular Coagulation (DIC), cerebral vascular accident, transient ischemic attack (TIA), acute coronary syndrome, or arterial systemic embolism.
7. Acute decompensated heart failure or cardiogenic shock at the time of randomization.
8. Severe sepsis or septic shock at the time of randomization.
9. The patient is a pregnant or lactating female.
10. Receipt of any of the following drugs or blood products within 7 days prior to consent:

    1. VKA (e.g., warfarin).
    2. Dabigatran.
    3. PCC (e.g., KCentra®) or rfVIIa (e.g., NovoSeven®), or anti-inhibitor coagulant complex (e.g., FEIBA®), FFP, and whole blood.
11. Past use of andexanet (or planned use of commercial andexanet).
12. Treatment with an investigational drug < 30 days prior to consent.
13. Any tumor-related bleeding.
14. Known hypersensitivity to any component of andexanet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (126):
- United States (10):
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Royal Oak, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Albany, New York
  - Research Site, Columbus, Ohio
  - Research Site, Tulsa, Oklahoma
  - Research Site, Allentown, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
- Austria (6):
  - Research Site, Innsbruck
  - Research Site, Klagenfurt
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Sankt Pölten
  - Research Site, Vienna
- Belgium (6):
  - Research Site, Belgium
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Ottignies
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, New Westminster, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Czechia (3):
  - Research Site, Brno
  - Research Site, Ostrava
  - Research Site, Prague
- Denmark (5):
  - Research Site, Aalborg
  - Research Site, Århus N
  - Research Site, Copenhagen
  - Research Site, Copenhagen Ø
  - Research Site, Odense C
- Finland (2):
  - Research Site, Helsinki
  - Research Site, Turku
- France (10):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Clermont-Ferrand
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Paris
  - Research Site, Suresnes
  - Research Site, Toulouse
- Germany (29):
  - Research Site, Altenburg
  - Research Site, Augsburg
  - Research Site, Bad Neustadt an der Saale
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Bremen
  - Research Site, Chemnitz
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Giessen
  - Research Site, Göttingen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Konstanz
  - Research Site, Lübeck
  - Research Site, Lünen
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Münster
  - Research Site, Osnabrück
  - Research Site, Sande
  - Research Site, Stuttgart
  - Research Site, Tübingen
  - Research Site, Ulm
- Greece (2):
  - Research Site, Alexandroupoli
  - Research Site, Athens
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Pécs
- Israel (6):
  - Research Site, Ashdod
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
- Italy (6):
  - Research Site, Bologna
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Perugia
  - Research Site, Roma
  - Research Site, Rome
- Research Site, Riga, Latvia
- Research Site, Vilnius, Lithuania
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Enschede
  - Research Site, Leiden
  - Research Site, Zwolle
- Research Site, Oslo, Norway
- Poland (3):
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Wejherowo
- Portugal (2):
  - Research Site, Coimbra
  - Research Site, Vila Nova de Gaia
- Russia (2):
  - Research Site, Arkhangelsk
  - Research Site, Novosibirsk
- Spain (7):
  - Research Site, Albacete
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (2):
  - Research Site, Lund
  - Research Site, Uppsala
- Research Site, Bern, Switzerland
- United Kingdom (6):
  - Research Site, Cambridge
  - Research Site, Harrow
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Eikelboom JW, Sharma M, Xu L, Bamberg K, Beyer-Westendorf J, Falkenberg C, Ladenvall P, Narayan R, Penland RC, Verhamme P, Shoamanesh A. Association of Biomarkers With Intracerebral Hematoma Expansion and Arterial Thromboembolic Events in Patients With Acute Intracranial Hemorrhage: The ANNEXA-I Biomarker Substudy. Stroke. 2025 Jul;56(7):1807-1815. doi: 10.1161/STROKEAHA.124.049966. Epub 2025 Apr 28. PMID 40289797
- [Derived] Shoamanesh A, Sharma M. Andexanet for Factor Xa Inhibitor-Associated Acute Intracerebral Hemorrhage. Reply. N Engl J Med. 2024 Aug 22;391(8):10.1056/NEJMc2407378#sa4. doi: 10.1056/NEJMc2407378. No abstract available. PMID 39167819
- [Derived] Connolly SJ, Sharma M, Cohen AT, Demchuk AM, Czlonkowska A, Lindgren AG, Molina CA, Bereczki D, Toni D, Seiffge DJ, Tanne D, Sandset EC, Tsivgoulis G, Christensen H, Beyer-Westendorf J, Coutinho JM, Crowther M, Verhamme P, Amarenco P, Roine RO, Mikulik R, Lemmens R, Veltkamp R, Middeldorp S, Robinson TG, Milling TJ Jr, Tedim-Cruz V, Lang W, Himmelmann A, Ladenvall P, Knutsson M, Ekholm E, Law A, Taylor A, Karyakina T, Xu L, Tsiplova K, Poli S, Kallmunzer B, Gumbinger C, Shoamanesh A; ANNEXA-I Investigators. Andexanet for Factor Xa Inhibitor-Associated Acute Intracerebral Hemorrhage. N Engl J Med. 2024 May 16;390(19):1745-1755. doi: 10.1056/NEJMoa2313040. PMID 38749032
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=18-513&attachmentIdentifier=86f20064-ee5c-4c94-9740-d31ff000e403&fileName=18-513-csr-study-synopsis_redacted_(1).pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data collected for the Andexanet Alfa arm were prespecified to be collected as a single Arm/Group regardless of the dose level the participant received.
Groups:
- Andexanet Alfa: Participants received a regimen of andexanet alfa administered as an intravenous (IV) bolus, immediately followed by a continuous infusion.
  Dosing regimen was based on which FXa inhibitor the participants received and the amount and timing of the most recent dose of treatment.
- Usual Care: Participants received usual care. Usual care consisted of any treatment(s) (including no treatment) other than andexanet alfa administered within 3 hours post-randomization that the Investigator and/or other treating physicians considered to be appropriate.
Period: Overall Study
Arm/Group | Andexanet Alfa | Usual Care
Started | 263 | 267
Received at Least 1 Dose of Study Drug | 262 | 265
Completed | 180 | 193
Not Completed | 83 | 74
Not completed — Death | 1 | 0
Not completed — Physician Decision | 3 | 1
Not completed — Other than Specified | 5 | 2
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Disease Progression | 8 | 13
Not completed — Adverse Event | 61 | 55

BASELINE CHARACTERISTICS:
Population: Measured in the Intent-to-Treat Population (ITT), Extended Population, which included all randomized participants according to the randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Andexanet Alfa | Usual Care | Total
Number analyzed (Participants) | 263 | 267 | 530
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.4 (8.51) | 78.7 (8.61) | 79.0 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 128 | 245
  Male | 146 | 139 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 13 | 28
  Not Hispanic or Latino | 227 | 237 | 464
  Unknown or Not Reported | 21 | 17 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 239 | 247 | 486
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Effective Hemostasis
Description: Effective hemostasis was defined as a change from baseline in National Institutes of Health Stroke Scale (NIHSS) of + 6 or less at the 12 hour timepoint and ≤35% increase in haematoma volume compared to baseline on a repeat computed tomography (CT) or magnetic resonance imaging (MRI) scan at 12 hours and no rescue therapies administered between 3 hours and 12 hours after randomization (defined as excellent or good hemostasis). The NIHSS is a validated quantitative assessment tool to measure stroke-related neurological deficits and ranges from 0 (no neurological deficits) to a maximum of 42, indicative of a very severe level of impairment. Data presented is for the number of participants who achieved effective hemostasis (excellent or good hemostasis), as adjudicated by the independent Endpoint Adjudication Committee (IEAC).
Time Frame: Baseline up to 12 hours
Population: Measured in the ITT set, primary efficacy population, which included all participants randomized to study intervention based on the first data cut-off. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Andexanet Alfa | Usual Care
Number analyzed (Participants) | 224 | 228
Participants | 150 | 121
Statistical Analysis 1: Comparison: Andexanet Alfa vs Usual Care; Test type: Other; p = 0.0032, Cochran-Mantel-Haenszel; Percentage proportion difference = 13.4, 95% CI 2-sided [4.6 to 22.2]

2. Secondary Outcome: Percentage Change From Baseline to Nadir in Anti-FXa Activity
Description: Anti-FXa activity was measured from plasma samples to assess the anticoagulant status of FXa inhibitors using a modified chromogenic assay performed at a Central Laboratory. Nadir was defined as the minimum anti-FXa activity post-randomization.
Time Frame: Baseline up to 2 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change
Arm/Group | Andexanet Alfa | Usual Care
Number analyzed (Participants) | 203 | 199
Percent change | -94.41 [-99.1 to 1805.0] | -27.46 [-97.9 to 416.0]
Statistical Analysis 1: Comparison: Andexanet Alfa vs Usual Care; Test type: Other; p < 0.0001, ANCOVA; Analysis presented for ANCOVA based on ranks; Difference in least squares mean = -185.99, 95% CI 2-sided [-199.93 to -172.05]

ADVERSE EVENTS:
Time Frame: Up to approximately 30 days
Description: All-cause mortality (ACM) is presented for all enrolled participants. Serious adverse events and other adverse event (AE) data are presented for all randomized participants who received study treatment and were analyzed according to the actual treatment received.
  ACM data includes participants who died due to AEs, an initial intracranial hemorrhage (disease progression), or participants who were discontinued from the study for other reasons and died on, or after, the day of discontinuation.
Arm/Group | Andexanet Alfa | Usual Care
All-Cause Mortality (participants affected / at risk) | 75/263 | 70/267
Serious Adverse Events (participants affected / at risk) | 120/262 | 96/265
Other Adverse Events (participants affected / at risk) | 198/262 | 200/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Andexanet Alfa (N=262) | Usual Care (N=265)
Myocardial infarction (Cardiac disorders) | 8 | 1
Acute myocardial infarction (Cardiac disorders) | 3 | 2
Cardiac failure (Cardiac disorders) | 3 | 0
Acute cardiac event (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac dysfunction (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Intestinal mass (Gastrointestinal disorders) | 0 | 1
Ischaemic enteritis (Gastrointestinal disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 14 | 16
Pneumonia aspiration (Infections and infestations) | 14 | 7
Sepsis (Infections and infestations) | 6 | 2
Urinary tract infection (Infections and infestations) | 4 | 1
Urosepsis (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 2
Brain herniation (Injury, poisoning and procedural complications) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 8 | 11
Cerebral haemorrhage (Nervous system disorders) | 7 | 11
Ischaemic stroke (Nervous system disorders) | 13 | 2
Hydrocephalus (Nervous system disorders) | 7 | 4
Neurological decompensation (Nervous system disorders) | 2 | 7
Cerebral haematoma (Nervous system disorders) | 3 | 5
Epilepsy (Nervous system disorders) | 1 | 2
Brain oedema (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebrospinal fluid circulation disorder (Nervous system disorders) | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cerebellar stroke (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebral vasoconstriction (Nervous system disorders) | 0 | 1
Cerebral venous thrombosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Intracranial haematoma (Nervous system disorders) | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Stroke in evolution (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Subdural hygroma (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 2 | 3
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary bladder rupture (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2
Haematoma (Vascular disorders) | 1 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Embolism arterial (Vascular disorders) | 1 | 0
Femoral artery embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Andexanet Alfa (N=262) | Usual Care (N=265)
Pneumonia (Infections and infestations) | 28 | 25
Pneumonia aspiration (Infections and infestations) | 19 | 16
Urinary tract infection (Infections and infestations) | 54 | 44
Hypokalaemia (Metabolism and nutrition disorders) | 40 | 28
Delirium (Psychiatric disorders) | 20 | 26
Insomnia (Psychiatric disorders) | 14 | 9
Headache (Nervous system disorders) | 24 | 19
Hypertension (Vascular disorders) | 18 | 19
Constipation (Gastrointestinal disorders) | 39 | 25
Nausea (Gastrointestinal disorders) | 23 | 17
Vomiting (Gastrointestinal disorders) | 9 | 14
Pyrexia (General disorders) | 23 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03661528/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT03661528/SAP_001.pdf